CLINICAL TRIAL: NCT01291589
Title: HIV Prevention in Very High Risk Men Who Have Sex With Men
Acronym: ENGAGE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: Massachusetts General Hospital (Other); Harvard University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Assistant Professor, Harvard Medical School, Director, Behavioral Medicine, Department of Psychiatry Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2P30AI060354-07 (NIH)
Record Dates: First submitted 2011-02-01; First posted 2011-02-08 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Risk Reduction Behavior
Keywords: HIV-infected; MSM; HIV prevention
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive-behavioral counseling (Experimental)
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Treatment will include elements from effective interventions for reducing risky sexual behaviors

SUMMARY:
The purpose of this study is to pilot test an innovative program development project in an open trial format an 8-session, individual, cognitive-behavioral therapy based, intervention on ten (10) HIV-infected men who have sex with men who report very high levels (>10 episodes) of sexual transmission risk behavior (unprotected anal intercourse with serodiscordant partners).

DETAILED DESCRIPTION:
This is an innovative program development project that will, over the next year, pilot test, in an open trial format an 8-session, individual, cognitive-behavioral therapy based, intervention on ten (10) HIV-infected men who have sex with men who report very high levels (>10 episodes) of sexual transmission risk behavior (unprotected anal intercourse with serodiscordant partners). That is, to pilot test a novel prevention intervention designed to effect reductions in sexual transmission risk behavior among the riskiest men in the largest HIV risk group in the US. Effecting even modest reductions in the mean number of risk acts in this group will likely have substantial public health significance through the number of averted new HIV infections. Traditional secondary HIV intervention strategies (e.g., Information, Motivation, Behavior change (IMB)) models only have modest effects for HIV-positive MSM and there is evidence to suggest that these effects tend to diminish over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Self-reports as a man who has sex with men (MSM)
* Self-reports being HIV-infected
* Reports engaging in 10 episodes or more of unprotected anal intercourse (receptive or insertive) in the past three months with male partners who are not HIV-infected or whose serostatus is unknown.
* Is capable of completing and fully understanding the informed consent process and the study procedures and assessments in English

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Decrease in self-reported sexual risk taking | Measured at baseline, 3 months post baseline (12 weeks) and again at 3 months post treatment (up to 24 weeks)
  The potential for an effect will determine the magnitude of the change in self-reported unprotected anal intercourse acts with HIV-uninfected and HIV-unknown status partners in the previous 3 months from baseline assessment to post treatment and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Conall M. O'Cleirigh, PhD, Principal Investigator — Fenway Community Health; Wade Taylor, PhD, Study Director — Fenway Community Health
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States